CLINICAL TRIAL: NCT04867694
Title: Impact Evaluation of a Package of Integrated and Multisectoral Services (PASIM) to Reduce Child Wasting in Chad
Brief Title: Integrated Research on Acute Malnutrition in Chad
Acronym: IRAM-CHAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: UNICEF (Other); Association Sahélienne de Recherches Appliquées pour le Développement Durable (Other); ONG Moustagbal (Unknown)
Responsible Party: Principal Investigator, Elodie Becquey, Senior Research Fellow, International Food Policy Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRAM-TCHAD
Record Dates: First submitted 2021-04-12; First posted 2021-04-30 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Acute Malnutrition in Childhood; Wasting
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Intervention Model Description: Non-blinded cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group receiving the standards of care and the usual activities of the partners without additional support from the IRAM project for the implementation of the PASIM. This includes the usual Community Management of Acute Malnutrition (CMAM) program. This group will also continue to benefit from the BCC and screening services already existing in their areas.
- Intervention (Experimental): The PASIM is delivered by the care groups. Each beneficiary is visited at home at least once a month (up to once a week if possible).
  The package of activities includes :
  Behavior change communication (all children in care groups)
  Monthly delivery of a nutritional supplement: limited to [6-11] months old children diagnosed as non-wasted (green MUAC) or for [6-59] months old for 6 months after discharge from the national CMAM program.
  Monthly delivery of a water purification input: limited to households with [6-11] months old children or with [6-59] months old children under CMAM treatment and for 6 months after discharge.
  Delivery of micronutrient powders to [12-23] months old children.
  Screening and referral for [6-59] months old children, formative supervision of MUAC measurement in families.
  Interventions: Behavioral: BCC; Dietary Supplement: Preventive supplement; Dietary Supplement: MNP; Other: Water purification input; Behavioral: Family MUAC; Behavioral: Screening by care group; Behavioral: CMAM compliance

INTERVENTIONS:
Behavioral: BCC — Behavior change communication on Nutrition, Health & Hygiene, including (but not limited to) awareness of dietary diversification from 6 months of age and adequate complementary feeding; and raising awareness of good water and hygiene practices.
  Arms: Intervention
Dietary Supplement: Preventive supplement — Monthly delivery of a nutritional supplement: enriched flour (CSB++), at a dose of 3 kg/month/beneficiary child. The nutritional supplement is limited to [6-11] months old children diagnosed as non-wasted (green MUAC); or children [12-59] months old for 6 months after discharge from a CMAM treatment or consolidation program.
  Arms: Intervention
Dietary Supplement: MNP — Delivery of micronutrient powders to [12-23] months old children (30 sachets per month for 2 months, every 6 months, according to international recommendations).
  Arms: Intervention
Other: Water purification input — Monthly delivery of a water purification input: bleach or flocculant/decontamination sachets for the potabilization of the water of the whole household. The water treatment input is limited to households with [6-11] months old children, or children [12-59] months old enrolled in a CMAM treatment program and for 6 months after discharge.
  Arms: Intervention
Behavioral: Family MUAC — One-time delivery of a mid-upper arm circumference (MUAC) measuring tape and training of families in its use, and actions to be taken based on the results. This will involve distributing Shakir bands to all households with [6-59] months old children and training mothers/guardians, or any other family members who express an interest, in screening for wasting using the MUAC criteria, and explaining the procedure to follow if the child tests positive in the family.
  Formative supervision of MUAC measurement in families. The training will be carried out by the members of the care groups and at each home visit, they will be able to ensure that the MUAC measurement technique is well mastered by the mother (or another member) and correct the technique if necessary.
  Arms: Intervention
Behavioral: Screening by care group — Monthly screening by the care group volunteers of the children they follow, using the MUAC.
  Referral to the health center of [6-59] months old children screened as malnourished (result of MUAC orange or red), and follow-up on referral to confirm child was enrolled
  Arms: Intervention
Behavioral: CMAM compliance — Weekly follow-up of [6-59] months old children under treatment and for 6 months after discharge from the national treatment and consolidation program : care group volunteers follow children under treatment until they recover and for the whole duration of their consolidation (for children cured of severe emaciation) through weekly home visits.
  They monitor treatment adherence (i.e., families follow the planned schedule of visits and receive inputs for treatment or consolidation) and treatment compliance (i.e., the malnourished or consolidating child receives the planned dose of therapeutic or supplementary food each day).
  Arms: Intervention

SUMMARY:
The IRAM Chad impact evaluation will be based on a cluster randomized controlled trial to study the impact of the integrated and multisectoral services package (PASIM), aimed at reducing the incidence and prevalence of wasting through integrated interventions, including, among other things, strengthening the activity of community care groups, food supplementation, water treatment, and screening for wasting conducted by families.

DETAILED DESCRIPTION:
The general objective of the integrated and multisectoral services package (PASIM) is to reduce the incidence and prevalence of wasting through integrated interventions, including, among other things, strengthening the activity of community care groups. The members of the care groups conduct home visits to children aged 6-23 months (or up to 59 months when the children are under treatment for wasting or have been discharged in the previous 6 months) to deliver messages for behavioral change related to complementary feeding, health and hygiene ; deliver nutritional supplement and water purification inputs; improve screening coverage (training and supervision of families to take the Mid-Upper Arm Circumference measurements, referral of malnourished cases); and verify adherence to treatment of malnourished cases, in the health district of Mongo, Guéra province, Chad, Central Africa.

The evaluation of the impact of PASIM will be based on a cluster randomized controlled trial, consisting of 100 villages or clusters of villages. The selected evaluation model will be that of a comparison of control groups (n=50; no implementation of the intervention) and intervention (n=50) through the follow-up of 3 cohorts :

1. Longitudinal in-home follow-up of a semi-open cohort of 1,750 children aged 6 months at enrollment (included continuously for 7 months and all followed through to the end of the study, which will last 9 months in total).
2. Longitudinal follow-up of all children aged 6-23 months enrolled for wasting treatment, based on health system records.
3. Longitudinal follow-up at home for 6 months of a closed cohort of 700 children aged 6-23 months at inclusion, discharged from a treatment for acute malnutrition.

The primary impact results are as follows:

* The longitudinal prevalence of wasting at the end of the study (Cohort 1).
* The recovery rate (Cohort 2).
* The incidence of relapse during the 11 months of the intervention (Cohort 3).

Secondary impact results include, but are not limited to :

* The incidence of wasting during the 11 months of the intervention (Cohort 1) ;
* The screening coverage (cohorts 1 and 3);
* The proportion of wasting cases enrolled in a treatment program (cohorts 1 and 3);
* The adherence to treatment (cohort 2) during the 11 months of the intervention.

ELIGIBILITY:
Cohort 1 (home visits):

The criteria for inclusion of children in the main cohort are:

* 6-6.9 months of age
* Child singleton
* The mother must live in the study area from the time of inclusion.
* The consent of the mother or guardian

The exclusion criteria are :

* Congenital malformations that make anthropometric measurements impossible.
* Mother intends to leave the study area by December 2021.

Cohort 2 (health registers-based):

The criteria for inclusion in the treatment cohort are :

* The child is included in a national treatment program.
* The child is between 6 and 23 months of age at inclusion
* Child lives in one of the 100 villages in the study area

Cohort 3 (home visits):

The inclusion criteria for the relapse study are:

* Child has been successfully treated for wasting (moderate or severe) and has been discharged from the national treatment program within the last 30 days.
* The child is between 6 and 23 months of age at inclusion.
* The child is singleton.
* The mother must live in the study area from the time of inclusion.
* The consent of the mother or guardian

The exclusion criteria are :

* Congenital malformations that make anthropometric measurements impossible.
* Mother intends to leave the study area by December 2021.

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2089 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Longitudinal prevalence of wasting among children enrolled at 6 months of age followed monthly until the end of the study (Cohort 1). | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  This indicator is defined for each child as the number of visits during which wasting is observed divided by the total number of monthly visits made (by interviewers).
Recovery rate in children enrolled at [6-23] months of age for up to 3 months of treatment and followed through to discharge (Cohort 2). | Up to 3 months, from date of inclusion in CMAM program until the date of recovery or 12th week after inclusion in CMAM program or date of death from any cause, whichever came first
  This indicator is defined as the number of discharges considered cured according to national program criteria (WHZ>-2 and MUAC>=125mm and absence of bilateral edema for two consecutive visits, within 12 weeks of enrollment in the program) divided by the total number of exits recorded.
Incidence of wasting in children enrolled at [6-23] months of age at discharge from a CMAM program cured, and followed for 6 months (Cohort 3). | Up to 6 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  This indicator is defined as the number of new cases of wasting recorded during monthly visits.

SECONDARY OUTCOMES:
Longitudinal prevalence of MAM (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  defined as the number of MAM diagnoses divided by the total number of monthly visits made
Longitudinal prevalence of SAM (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  Defined as the number of SAM diagnoses divided by the total number of monthly visits made
Incidence of wasting, MAM and SAM (cohort 1) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  defined as the number of new cases of wasting, MAM and SAM recorded during monthly visits among children enrolled at 6 months of age followed monthly until the end of the study (Cohort 1).
Incidence of MAM and SAM (cohort 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  defined as the number of new cases of MAM and SAM recorded during monthly visits.
prevalence of anemia (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression
  Proportion of children with a hemoglobin level below 11g/dl
Mean hemoglobin concentration (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression
  Mean hemoglobin concentration measures by hemocue reader
Prevalence of stunting (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  proportion of children with HAZ <-2 (relative to the 2006 WHO reference)
Height-for-age Z-score (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  Height-for-age Z-score relative to the 2006 WHO reference
Longitudinal wasting screening coverage (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  defined as the proportion of children screened (using MUAC, weight-for-height or bilateral edema) in the month prior to the monthly visit. Two sub-outcomes will also be concerned:
  * Screening coverage by care groups.
  * Coverage of the family MUAC component, which is the screening performed by a family member in the past month.
Referral rate of positive screenings (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  defined as the proportion of children who tested positive during the month (according to the mother) and not under CMAM treatment who were referred to the health center or FARNE site.
Enrollment of wasting, MAM, and SAM cases (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  proportion of cases who tested positive in the month prior to the monthly visit and not under CMAM treatment who were enrolled in a CMAM treatment program.
Linear growth rate (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  change in height-for-age index per month
Speed of weight growth (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  change in weight-for-height index per month
Weight gain (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  weight change per month
MUAC gain (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  change in MUAC per month
longitudinal prevalence of childhood morbidity, i.e. acute respiratory infections, fever, diarrhea and malaria (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  the number of diagnoses of daily signs of these morbidities divided by the total number of days reported (1-3 per monthly visit made).
Parental knowledge of nutrition, WASH, and health best practices (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  expressed as cumulative total and domain scores
Longitudinal prevalence of minimum dietary diversity of infant and young children (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  the proportion of children who consumed at least 5 of the 8 food groups (including breast milk) the day before the survey.
Longitudinal prevalence of Introduction of (semi) solid and soft complementary foods (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  the proportion of children 6-8 months of age who consumed (semi) solid and soft complementary foods the day before the survey Minimum dietary diversity in children, defined as the proportion of children who consumed at least 5 of the 8 food groups (including breast milk) the day before the survey.
  Minimum meal frequency for children, defined as the proportion of children who had eaten the day before the survey: 2 meals for breastfed children 6-8 months, 3 meals for breastfed children 9-23 months, or 4 meals for non-breastfed children 6-23 months.
  Minimum acceptable diet, defined as the proportion of children with both minimal dietary diversity and minimal meal frequency on the day before the survey.
  Consumption of iron-rich or iron-fortified foods in children.
Longitudinal prevalence of minimum meal frequency (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  the proportion of children who consumed the minimum recommended number of meals for their age on the day before the survey Minimum dietary diversity in children, defined as the proportion of children who consumed at least 5 of the 8 food groups (including breast milk) the day before the survey.
  Minimum meal frequency for children, defined as the proportion of children who had eaten the day before the survey: 2 meals for breastfed children 6-8 months, 3 meals for breastfed children 9-23 months, or 4 meals for non-breastfed children 6-23 months.
  Minimum acceptable diet, defined as the proportion of children with both minimal dietary diversity and minimal meal frequency on the day before the survey.
  Consumption of iron-rich or iron-fortified foods in children.
Practices related to water, hygiene and sanitation (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  Standard USAID indicators related to drinking water source, treatment, storage; hand washing; and sanitation
Vaccination coverage (cohorts 1 & 3) | Up to 9 months, from date of enrolment until the date of last documented progression or date of death from any cause, whichever came first
  Proportion of children with complete vaccination for their age
weight-for-height in z-score at enrollment in CMAM (cohort 2) | at the date of inclusion in CMAM program
  weight-for-height in z-score (relative to the 2006 WHO reference)
MUAC at enrollment in CMAM (cohort 2) | at the date of inclusion in CMAM program
  Mid-upper arm circumference (mm)
Duration of CMAM treatment (cohort 2) | Up to 3 months, from date of inclusion in CMAM program until the date of recovery or 12th week after inclusion in CMAM program or date of death from any cause, whichever came first
  defined as the number of days spent on treatment (enrollment and discharge) in children 6-23 months of age at enrollment, according to health registers
Treatment adherence (cohort 2) | Up to 3 months, from date of inclusion in CMAM program until the date of recovery or 12th week after inclusion in CMAM program or date of death from any cause, whichever came first
  defined as the proportion of cases enrolled for treatment who received timely treatment from dedicated services until recovery
Treatment outcomes (drop-out, death, transfer, non-response rates) (cohort 2) | Up to 3 months, from date of inclusion in CMAM program until the date of recovery or 12th week after inclusion in CMAM program or date of death from any cause, whichever came first
  Among proportion of cases enrolled for treatment
longitudinal prevalence of childhood morbidity (cohort 2) | Up to 3 months, from date of inclusion in CMAM program until the date of recovery or 12th week after inclusion in CMAM program or date of death from any cause, whichever came first
  defined by the number of days for which signs of these morbidities were reported divided by the total number of days observed/reported in the recall periods.

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Huybregts, PhD, Principal Investigator — IFPRI; Elodie Becquey, PhD, Principal Investigator — IFPRI; Jef Leroy, PhD, Principal Investigator — IFPRI
Locations (1):
- Mongo Health District, Mongo, Guéra Region, Chad

IPD SHARING:
Plan to Share IPD: Yes
In accordance with IFPRI's policy on research data management and open access, at the time of publication of scientific articles presenting results, the fully anonymized databases will become a public good and will be made available to the scientific community, government, and partners.
Supporting Information: Study Protocol, SAP
Time Frame: at the time of publication of scientific articles presenting results, the fully anonymized databases will become a public good and will be made available to the scientific community, government, and partners.

DOCUMENTS (2):
  • Study Protocol (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/94/NCT04867694/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT04867694/SAP_001.pdf